CLINICAL TRIAL: NCT05271656
Title: Evaluation of C-Scan Capsule in Identifying Subjects With Elevated Risk of Colon Polyps
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Check Cap board of directors decision to stop all company activities including clinical trails
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL-SY-02-0100
Record Dates: First submitted 2022-02-15; First posted 2022-03-09 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Masking Description: The Sponsor and the C-Scan data analysis team shall be blind to subject's optical colonoscopy data until the C-Scan report is created.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- C-Scan System (Experimental): All study participants will undergo the C-Scan System procedure, followed by a standard of care optical colonoscopy
  Interventions: Device: C-Scan System

INTERVENTIONS:
Device: C-Scan System — Subjects will be provided with contrast agent and dietary fiber pills, and instructed to start intake of fiber pills 5 days, and contrast agent 48 hours prior to scheduled C-Scan capsule ingestion. C-Scan system intervention includes ingestion of the C-Scan Cap and attachment of the C-Scan Track to the subject's lower back. The subject is required to keep the C-Scan Track attached to the lower back and to continue intake of contrast agent and dietary fiber pills until the C-Scan Cap's natural excretion. Standard of care optical colonoscopy will be performed within 60 days from the C-Scan Cap ingestion.
  Other Names: Optical colonoscopy

SUMMARY:
The main objective of the study is to determine the ability of the C-Scan system to identify subjects who are at elevated risk for colon polyps. This will be evaluated by comparing the C-Scan data to colonoscopy data. The C-Scan procedure is therefore performed before the colonoscopy procedure, in order to compare these tests and evaluate the C-Scan system's effectiveness.

During the C-scan procedure, Subjects will be asked to come for an appointment in a clinic, during this appointment, the C-Scan Track will be placed on the participant's back. The participant will then be asked to swallow the C-Scan capsule whereafter they are free to continue their routine. Participants will start intake of fiber pills 5 days, and contrast agent 48 hours prior to C-Scan capsule ingestion and will continue intake up to the capsule's natural excretion.

A standard colonoscopy procedure will be performed within 60 days following C-Scan Cap ingestion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 45-75 years old
2. Able to provide a signed informed consent.
3. Willing and able to comply with the specified study requirements and can be contacted by telephone.
4. Scheduled for colonoscopy procedure no later than 60 days after C-Scan ingestion
5. Maximal abdominal circumference < 125 cm.

Exclusion Criteria:

1. Subject who is not a suitable candidate for a colonoscopy
2. Known history of dysphagia or other swallowing disorders.
3. History of the following:

   1. Colorectal polyps
   2. A personal history of CRC
   3. A family history of CRC or adenomatous polyps diagnosed in a relative before 60 years of age
   4. A history of inflammatory bowel disease of significant duration
   5. One of two (2) hereditary syndromes
4. Known motility disorders:

   1. Chronic Constipation: less than three (3) bowel movements/week, without the use of laxatives within the last 3 months.
   2. Ongoing diarrhea defined as passage of loose or watery stools at least three times within 24-hour
   3. Delayed gastric emptying.
5. Known IBD (Crohn's, Ulcerative Colitis)
6. Prior history of gastrointestinal tract surgery.
7. Prior history of abdominal surgery that might cause bowel strictures leading to capsule retention, as determined by a physician
8. Any condition believed to have an increased risk for capsule retention, known strictures, known bowel adhesion or 'obstacles' to free passage of the capsule (such as esophageal diverticulosis, intestinal tumors, radiation enteritis) or incomplete colonoscopies as determined by a physician.
9. Significant change in diameter and frequency of stool within the last 3 months.
10. GI bleeding within the last 3 months i.e., rectal outlet bleeding, hematochezia or melena.
11. Implanted cardiac device or any other implanted active device
12. Known sensitivity to iodine
13. Acute kidney failure
14. Known condition which precludes compliance or is contraindicated with study and/or device instructions.
15. Any procedure requiring contrast agent, or which may introduce electronic interference (such as magnetic resonance imaging, DEXA scan) or an imaging procedure pre-scheduled within 14 days of C-Scan ingestion
16. Nuclear imaging procedure within the four (4) weeks preceding the C-Scan procedure.
17. Known condition of opioid use disorder and/or alcoholism.
18. Women who are either pregnant or nursing at the time of screening (to be verified by urine or serum pregnancy test for woman of child- bearing potential who are not post-menopausal or undergone surgical sterilization).
19. Concurrent participation in another clinical trail using any investigational drug or device.
20. Previous colonoscopy performed five (5) years or less before date of enrolment
21. Subjects who tend to hyperhidrosis in the back area

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Demonstrate the accuracy of the C-Scan system in identifying subjects with colon polyps comparing to optical colonoscopy (OC). | 60 days
  For each subject the primary efficacy endpoints are dichotomous diagnosis using the C-Scan device (Test) and optical colonoscopy (Reference standard).
  Reference standard will be considered "positive" ("1") if at least one polyp of at least 6 mm is found.
  Test will be considered with elevated risk for polyps ("1") if either at least one polyp of at least 6 mm is found or long WGTT* occurred.
  The above endpoints will be used to calculate sensitivity and specificity examined in the primary analysis.
  *Long WGTT is defined as more than 73 hours for male and more than 97 hours for female.

SECONDARY OUTCOMES:
Negative predictive value for ruling out polyps of at least 10 mm. | 60 days
  Reference standard will be considered "positive" ("1") if at least one polyp of at least 10 mm is found.
Sensitivity of C-Scan for detecting polyps of at least 10mm. | 60 days
  Reference standard will be considered "positive" ("1") if at least one polyp of at least 10 mm is found.
Demonstrate the safety of the C-Scan System | 7±3 days from capsule excretion
  Frequency of patients who experienced device or procedure related serious adverse events up to 7±3 days from capsule excretion. In addition, AEs and SAEs will be presented by severity and relation to device and procedure.
Demonstrate subjects' satisfaction and usability with the C-Scan System | 7±3 days from capsule excretion
  This will be assessed via a descriptive analysis using a questionnaire
Demonstrate subjects' satisfaction with the C-Scan System compared to optical colonoscopy | 4-10 days post colonoscopy
  This will be assessed via a descriptive analysis using a questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided